CLINICAL TRIAL: NCT05258123
Title: The Effects of Ginkgo Biloba Extract in the Treatment of Schizophrenia
Brief Title: Ginkgo Biloba Extract in the Treatment of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Professor, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CASPsy4
Record Dates: First submitted 2022-02-24; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; Ginkgo biloba extract; cognition
MeSH Terms: conditions — Schizophrenia | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active drug (Active Comparator): A fixed titration to 360mg （or nine tables） daily of Ginkgo biloba extract was administered with three times daily dosage throughout the study
  Interventions: Drug: Ginkgo Biloba Extract
- placebo (Placebo Comparator): A nine tables of placebo were administered with three times daily dosage throughout the study
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Ginkgo Biloba Extract — Ginkgo biloba extract with 360mg was administered
  Arms: active drug
Drug: Placebo oral tablet — Placebo with nine tables was administered
  Arms: placebo

SUMMARY:
We investigated the effects of Ginkgo biloba extract on the symptoms and cognitive functioning in patients with schizophrenia

DETAILED DESCRIPTION:
Objective: This study aimed to evaluate the effect of Ginkgo biloba extract in the treatment of symptoms and cognitive functioning in 200? chronic patients with schizophrenia

Methods:

1. Clinical Trial: This is a randomized, double-blind and parallel controlled trial in the chronic patients with schizophrenia. The study consists of 12 weeks of double-blind treatment.
2. Assessment Procedures:

2.1 Primary Outcome Variable: Patients were assessed by two clinical trained staff, who were blind to the treatment protocols, by using the Positive and Negative Syndrome Scale (PANSS) to assess the psychopathology and Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) to evaluation the cognitive functioning. Patients were interviewed at screening, and at baseline, 4? weeks, 12? weeks.

2.2 Side effects: The side effect rating scale (UKU) was used to assess the side effect at baseline, 4? weeks, and 12? weeks.

2.3 Weight gain measurement: weigh was measured every week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia by two senior psychiatrists
* Between 18 and 60 years and Han Chinese
* Duration of symptoms at least 12 months
* Current psychotic symptoms of moderate severity

Exclusion Criteria:

* A Diagnostic and Statistical Manual of Mental Disorders IV Axis I diagnosis other than schizophrenia
* Documented disease of physical diseases including, but not limited to stroke, tumor, Parkinson's disease, Huntington's disease, seizure, epilepsy, history of brain trauma；
* Pregnant or breast-feeding female'
* Subjects who suffered from alcohol or illegal durg abuse/dependence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
clinical symptoms | 12 weeks
  symptoms assessed on PANSS
cognitive functioning | 12 weeks
  cognitive functioning assessed on RBANS

SECONDARY OUTCOMES:
Side effects | 12 weeks
  side effect assessed on UKU

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Y Zhang, M.D, Ph.D, Principal Investigator — Institute of Psychology, Chinese Academy of Sciences
Locations (1):
- Beijing HuiLongGuan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Data with be available on request

REFERENCES:
- [Background] Montes P, Ruiz-Sanchez E, Rojas C, Rojas P. Ginkgo biloba Extract 761: A Review of Basic Studies and Potential Clinical Use in Psychiatric Disorders. CNS Neurol Disord Drug Targets. 2015;14(1):132-49. doi: 10.2174/1871527314666150202151440. PMID 25642989
- [Background] Zheng W, Xiang YQ, Ng CH, Ungvari GS, Chiu HF, Xiang YT. Extract of Ginkgo biloba for Tardive Dyskinesia: Meta-analysis of Randomized Controlled Trials. Pharmacopsychiatry. 2016 May;49(3):107-11. doi: 10.1055/s-0042-102884. Epub 2016 Mar 15. PMID 26979525
- [Background] Zhang WF, Tan YL, Zhang XY, Chan RC, Wu HR, Zhou DF. Extract of Ginkgo biloba treatment for tardive dyskinesia in schizophrenia: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2011 May;72(5):615-21. doi: 10.4088/JCP.09m05125yel. Epub 2010 Sep 21. PMID 20868638